CLINICAL TRIAL: NCT00268151
Title: Phase I Study of Oxaliplatin (Eloxatin) and Capecitabine (Xeloda) and Concurrent Radiation Therapy (XELOX-RT) in Non-Small Cell Lung Cancer
Brief Title: Oxaliplatin in Combination With Capecitabine and Concurrent Radiation Therapy in Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to lack of funding.
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other); Sanofi (Industry)
Responsible Party: Principal Investigator, Goetz Kloecker, Associate Professor, University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 562.04; OX-03-156
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: non-small cell lung cancer; oxaliplatin; capecitabine; XELOX-RT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Oxaliplatin; Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin
Drug: Capecitabine

SUMMARY:
The purpose of this study is to determine the most suitable dose of Oxaliplatin that can be safely given in combination with a low fixed dose of Capecitabine and a limited volume of radiation in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
The purpose of this study is to determine the maximum tolerated dose (MTD) and the dose limiting toxicity (DLT) of Oxaliplatin in combination with Capecitabine and radiation in subjects with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven non-small cell lung cancer
* inoperable Stage III A or B NSCLC
* must have measurable disease by RECIST criteria
* no more than one prior chemotherapy for advanced disease
* ECOG Performance Status of 0, 1, or 2
* must be able to swallow pills or have a working gastric feeding tube and no evidence of malabsorption
* negative serum beta-HCG test and under active contraception (for females of childbearing potential)
* no known allergies to any of the study drugs
* willingness to sign an informed consent

Exclusion Criteria:

* women who are pregnant or breastfeeding
* ANC of less than 1500/mm3
* platelet count of less than 100,000/mm3
* estimated creatinine clearance of less than 50 cc/min (as measured by the Cockcroft-Gault equation)
* bilirubin of less than 2mg/dl
* SGPT of greater than 2x nl
* peripheral neuropathy of Grade 2 or higher
* more than one previous chemotherapy and previous radiation therapy to the chest
* a history of CHF/MI or other significant cardiac history within the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-02; Primary Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Goetz H Kloecker, MD, MSPH, Principal Investigator — James Graham Brown Cancer Center/ University of Louisville
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

REFERENCES:
- See also: James Graham Brown Cancer Center — http://www.browncancercenter.org